CLINICAL TRIAL: NCT05290753
Title: Impact of Prokinetic Use After Emergency Intestinal Anastomosis on Short and long_term Clinical Outcome
Brief Title: Impact of Prokinetic Use After Emergency Intestinal Anastomosis on Postoperative Clinical Outcomes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Doha Adel Noureldin, Resident doctor at general surgery department sohag university hospital, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Soh-Med-22-02-09
Record Dates: First submitted 2022-03-04; First posted 2022-03-22 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: Prokinetic Use After Emergency Intestinal Anastomosis
MeSH Terms: interventions — Erythromycin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prokinetic use in accelerate healing of urgent intestinal anastomosis (Other): Prikinetic agents administered immediately post operative and time of stay at hospital twice daily
  Interventions: Drug: Prokinetic Motility Agents as primpiram and gastreg

INTERVENTIONS:
Drug: Prokinetic Motility Agents as primpiram and gastreg — Prospective cohort study to evaluate the effect of pro kinetic use in emergency intestinal anastomosis
  Other Names: Primpiram and gastreg and erythromycin

SUMMARY:
Prokinetic drugs used to accelerate healing of intestinal anastomosis of urgent cases which not prepared preoperative by increase intestinal motility and gastric emptying and decrease postoperative adhesions They are many types of prokinetics as cholinergic agonists, dopamine antagonist, serotonergic agonists and macrolides Agents of prokinetics administered immediately post operation and at the time of hospitalization

DETAILED DESCRIPTION:
By evaluation the effect of prokinetic use versus non use after emergency intestinal intestinal anastomosis on short and long term clinical outcome It will be prospective cohort study which conducted in sohag university hospital Study will include patients presented with urgent anastomosis Inclusion criteria: all adults underwent emergency intestinal anastomosis Exclusion criteria: pediatrics, patients with comorbidities and patients with electively resection and anastomosis.

Primary goals are to detect effect of prokinetics on incidence of leakage rate Secondary outcomes include early bowel opening, enteral feeding, post operative pain, wound infection and adhesion formation rate.

ELIGIBILITY:
Inclusion Criteria:

* all adult patients

Exclusion Criteria:

* pediatrics
* patients associated with comorbidities
* patients with electively resection and anastomosis

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Leakage rate | 5 days postoperative
  Fecal fistula

SECONDARY OUTCOMES:
Early bowel opening | 3 days postoperative
  Duration taken to patient to pass feces and flatus

CONTACTS AND LOCATIONS:
Overall Officials: Alaa eldin Hassan, Professor, Study Director — Professor of general surgery
Locations (1):
- Of medicine, Sohag university hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Evaluate the use of prokinetic versus non use in emergency intestinal anastomosis
Supporting Information: Study Protocol
Time Frame: 6 months
Access Criteria: Evaluate effect of use of pro kinetic drug versus non use in emergency intestinal analstomosis

REFERENCES:
- [Background] Acosta A, Camilleri M. Prokinetics in gastroparesis. Gastroenterol Clin North Am. 2015 Mar;44(1):97-111. doi: 10.1016/j.gtc.2014.11.008. Epub 2014 Dec 23. PMID 25667026